CLINICAL TRIAL: NCT05554471
Title: A Multicenter, Prospective, Randomized, Controlled, Open Label Trial to Evaluate the Safety and Efficacy of Mynx Control Venous Vascular Closure Device 6F-12F vs Manual Compression in Patients Who Have Undergone Endovascular Procedures Utilizing up to 12F Procedural Sheaths
Brief Title: Evaluation of Safety and Efficacy of the Mynx Control Venous Vascular Closure Device 6F-12F vs Manual Compression
Acronym: ReliaSeal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P22-8301
Record Dates: First submitted 2022-09-20; First posted 2022-09-26 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Venous Vascular Closure
Keywords: manual compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Mynx Control Venous Closure (Experimental): 204 (2:1 randomized - 136 VCD:68 manual compression)
  Interventions: Device: MYNX CONTROL™ Venous Vascular Closure Device 6F-12F
- Manual Compression (Active Comparator): 204 (2:1 randomized - 136 VCD:68 manual compression)
  Interventions: Device: MYNX CONTROL™ Venous Vascular Closure Device 6F-12F

INTERVENTIONS:
Device: MYNX CONTROL™ Venous Vascular Closure Device 6F-12F — Mynx Control Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation.

SUMMARY:
ReliaSeal is a clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs.

DETAILED DESCRIPTION:
ReliaSeal is a multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. The study is planned to enroll 204 patients with an additional group of patients to be part of the initial roll-in phase. Up to two (2) roll-in patients per physician will be allowed. All patients who sign the informed consent and randomized to either treatment arm will be followed through 30 days post procedure. There will be up to 15 participating study sites, with a minimum of five (5) sites, all located in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Able and willing to provide informed consent and to complete a follow-up visit at 30 days
3. Planned catheter-based procedures via the common femoral vein(s) using up 6F to 12F introducer sheaths which meet indications for elective, nonemergent interventions of disease state, without contraindications for emergent vascular surgery or manual compression of the venous access sites

Exclusion Criteria:

1. Any use of systemic steroids (IV or oral) within 30 days of procedure
2. History of deep vein thrombosis, pulmonary embolism, or thrombophlebitis within 6 months of procedure
3. Presence of thrombocytopenia (platelet count < 100,000 cells/mm3) or anemia (hemoglobin < 10 g/dL, hematocrit < 30%)
4. History of bleeding disorders such hemophilia or von Willebrand's disease
5. Currently involved in any other investigational clinical trial
6. Documented history of uncontrolled hypertension (i.e., systolic blood pressure > 180 mm Hg), or critical illness requiring intravenous vasopressors for blood pressure stabilization
7. Femoral arteriotomy or venotomy in either limb within 10 days pre procedure
8. Use of VCD in either limb within 30 days of procedure
9. Any planned procedure involving femoral arterial or venous access in either limb within 30 days or prior to study exit
10. Renal insufficiency (i.e., serum creatinine > 2.5 mg/dL)
11. Patients who are pregnant, planning to become pregnant during the study period, or lactating
12. Body-mass index (BMI) > 45 kg/m2 or <20 kg/m2
13. Unable to routinely walk at least 20 feet without assistance
14. Known allergy/adverse reaction to polyethylene glycol or contrast medium
15. Planned procedures (including staged) or concomitant conditions/comorbidities that per investigator's judgment may extend ambulation attempts beyond 2-3 hours, and/or require extended hospitalization or re-hospitalization
16. Previous vascular surgery or repair in the vicinity of the target access site within the previous 90 days of the procedure
17. Active systemic infection, or cutaneous infection or inflammation in the vicinity of the target access site
18. Current COVID-19 infection (with or without symptoms), positive test for COVID- 19 within 14 days, or recent exposure to a person with COVID-19 infection
19. Patients who refuse blood transfusion if it were to be needed
20. Patients with expected life of less than 30 days

Intra-Procedural Exclusion Criteria

Patients who meet any of the following criteria during the index procedure will be excluded:

1. Any attempt at femoral arterial access or inadvertent arterial puncture with hematoma during the procedure
2. Any procedural complications that may interfere with routine recovery, ambulation, or discharge eligibility times
3. Physician deems that a different hemostasis approach for venous access sites is necessary
4. Physician deems that the subject should not attempt protocol required ambulation (reference ambulation protocol per section 14.2)
5. Venous access site location is noted to be above the inguinal ligament (cephalad to lower half of the femoral head or the inferior epigastric vein origin from the external iliac vein)
6. Intra-procedural bleeding around sheath, or suspected intraluminal thrombus, hematoma, pseudoaneurysm, or AV fistula
7. Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, accidental arterial stick with hematoma, "back wall stick", etc.)
8. A < 6F or > 12F procedural sheath is present at any time during the procedure or at closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Colorado Heart and Vascular PC, Lakewood, Colorado
  - Baptist Health Miami Cardiac and Vascular Institute, Miami, Florida
  - Palm Vascular Centers, Miami Beach, Florida
  - Tampa Cardiovascular Interventions and Research, Tampa, Florida
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Hightower Clinical, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - OnSite Clinical Solutions, Rock Hill, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Rio Grande Regional Hospital, McAllen, Texas
  - North Dallas Research Associates, McKinney, Texas

REFERENCES:
- [Result] Summers J, Swarup V, Parker I, Bumgarner J, Brenyo A, Saleh L, Sadanandan S, Sanchez J, Beasley R, Gupta S; other members of the ReliaSeal Study Group. Safety and Efficacy of a Novel Sealant-Based Vascular Closure Device Following Electrophysiology Procedures: ReliaSeal Trial. J Cardiovasc Electrophysiol. 2025 May;36(5):1022-1031. doi: 10.1111/jce.16623. Epub 2025 Mar 17. PMID 40098328
- See also: Original Article, First published: 17 March 2025 — http://onlinelibrary.wiley.com/doi/10.1111/jce.16623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began on 30Aug2022, and enrollment ended on 22May2023.
Pre-assignment Details: 352 subjects agreed to participate in the study following the completion of the informed consent process. Among 352 enrolled subjects, 44 were included as roll-in subjects, and 38 were screen failures. Both roll-in and screen-failed subjects were not assigned to either arm.
Groups:
- MYNX CONTROL™ VENOUS VCD: Patients received MYNX CONTROL™ Venous Vascular Closure Device 6F-12F in sealing femoral venous access sites. The patients have undergone endovascular procedures utilizing one or more procedural sheaths up to 12F.
- Manual Compression: Patients received Manual Compression in sealing femoral venous access sites. The patients have undergone endovascular procedures utilizing one or more procedural sheaths up to 12F.
Period: Overall Study
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
Started | 177 | 93
Completed | 173 | 90
Not Completed | 4 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Manual Compression: Patients received Manual Compression in sealing femoral venous access sites.The patients have undergone endovascular procedures utilizing one or more procedural sheaths up to 12F.
- Total: Total of all reporting groups
Arm/Group | MYNX CONTROL™ Venous VCD | Manual Compression | Total
Number analyzed (Participants) | 177 | 93 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 26 | 87
  >=65 years | 116 | 67 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (11.62) | 66.8 (10.63) | 66.7 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 32 | 92
  Male | 117 | 61 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 2 | 11
  Not Hispanic or Latino | 158 | 87 | 245
  Unknown or Not Reported | 10 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 167 | 89 | 256
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 177 | 93 | 270

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Major Complications of the Target Limb Access Site Within 30 Days
Description: Defined as the rate of CEC adjudicated combined major venous access site closure-related complications through 30 days post-procedure, attributed directly to VCD or Manual Compression without other likely cause.
Time Frame: 30 days post procedure
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
Number analyzed (Participants) | 177 | 93
Number analyzed (limbs) | 229 | 119
limbs | 0 | 1

2. Primary Outcome: Primary Effectiveness Endpoint: Time to Ambulation
Description: Defined as time (in hours) between removal of the MYNX CONTROL™ Venous Vascular Closure Device 6F-12F device (device group) or of the final sheath (control group) and when subject stands and walks 20 feet without evidence of rebleeding from any femoral venous access site.
Time Frame: Post procedure
Population: Five (5) MYNX CONTROL VENOUS VCD subjects with missing data and Two (2) Manual Compression subjects with missing data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
Number analyzed (Participants) | 172 | 91
hours | 2.6 (1.03) | 5.1 (4.35)
Statistical Analysis 1: Comparison: MYNX CONTROL™ VENOUS VCD vs Manual Compression; Hypothesis: the time to ambulation for the subjects using the MYNX CONTROL™ Venous VCD was significantly less than for those where manual compression was used; Test type: Superiority; p < 0.001, t-test, 1 sided

3. Primary Outcome: Primary Effectiveness Endpoint: Time to Hemostasis
Description: Defined as time (in minutes) between removal of each MYNX CONTROL™ Venous Vascular Closure Device 6F-12F device (device group) or of each sheath (control group) and first observed and confirmed venous hemostasis (per access site analysis).
Time Frame: Post procedure
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: access sites
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
Number analyzed (Participants) | 177 | 93
Number analyzed (access sites) | 470 | 249
minutes | 2.1 (1.79) | 11.4 (7.19)
Statistical Analysis 1: Comparison: MYNX CONTROL™ VENOUS VCD vs Manual Compression; Hypothesis: the time to hemostasis for the MYNX CONTROL™ Venous VCD device is at least 5 minutes less than manual compression; Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: Secondary Safety Endpoints: Minor Complications of the Target Limb Access Site Within 30 Days
Description: Defined as the rate of CEC adjudicated combined minor venous access site closure-related complications through 30 days post-procedure, attributed directly to MYNX CONTROL™ Venous VCD or Manual Compression without other likely cause.
Time Frame: 30 days post procedure
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
Number analyzed (Participants) | 177 | 93
Number analyzed (limbs) | 229 | 119
limbs | 0 | 6

5. Secondary Outcome: Time to Discharge Eligibility
Description: Defined as elapsed time (in hours) between removal of the final MYNX CONTROL™ Venous VCD or removal of the final sheath and when subject is eligible for discharge from the institution based on the assessment of the attending physician.
Time Frame: Post Procedure
Population: There were 4 missing data in the MYNX CONTROL VENOUS VCD group and 2 missing data in the Manual Compression group
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
Number analyzed (Participants) | 173 | 91
hours | 3.1 (1.24) | 5.5 (4.58)
Statistical Analysis 1: Comparison: MYNX CONTROL™ VENOUS VCD vs Manual Compression; Hypothesis: The time to discharge eligibility for the subjects using the MYNX CONTROL™ Venous VCD was significantly less than for those where manual compression was used; Test type: Superiority; p < 0.001, t-test, 1 sided

6. Secondary Outcome: Procedural Success
Description: Defined as attainment of final hemostasis at all venous access sites without major venous access site closure-related complications through 30 days.
Time Frame: 30 days post procedure
Population: Six (6) MYNX CONTROL VENOUS VCD subjects with missing data and three (3) Manual Compression subjects with missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
Number analyzed (Participants) | 171 | 90
Participants | 171 | 89

7. Secondary Outcome: Device Success
Description: Defined as the ability to successfully deploy the MYNX CONTROL™ VENOUS VCD delivery system, deliver the polyethylene glycol hydrogel sealant, and achieve hemostasis.
Time Frame: During procedure
Measure: Count of Units; unit: access sites
Units Other Than Participants: access sites
Arm/Group | MYNX CONTROL™ VENOUS VCD
Number analyzed (Participants) | 177
Number analyzed (access sites) | 470
access sites | 470

ADVERSE EVENTS:
Time Frame: 30 days follow-up
Description: Two (2) MYNX CONTROL VENOUS VCD subjects and one (1) Manual Compression subject were terminated prior to the procedure and were missing data.
Arm/Group | MYNX CONTROL™ VENOUS VCD | Manual Compression
All-Cause Mortality (participants affected / at risk) | 0/175 | 1/92
Serious Adverse Events (participants affected / at risk) | 10/175 | 4/92
Other Adverse Events (participants affected / at risk) | 16/175 | 5/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MYNX CONTROL™ VENOUS VCD (N=175) | Manual Compression (N=92)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Psychogenic seizure (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Vascular compression (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MYNX CONTROL™ VENOUS VCD (N=175) | Manual Compression (N=92)
Procedural nausea (Injury, poisoning and procedural complications) | 11 | 0
Haematoma (Vascular disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT05554471/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT05554471/SAP_001.pdf